CLINICAL TRIAL: NCT04186065
Title: Cross-Sectional Study: The Prevalence of White Spot Lesions During Orthodontic Treatment With Fixed Appliances
Brief Title: The Prevalence of White Spot Lesions During Orthodontic Treatment With Fixed Appliances
Acronym: WSLs
Status: Completed | Type: Observational
Sponsor: Hiroko Nagaoka (Other)
Responsible Party: Sponsor-Investigator, Hiroko Nagaoka, Special Faculty, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 47148
Record Dates: First submitted 2019-06-24; First posted 2019-12-04 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Dental Caries
Keywords: white spot; lesions; tooth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates how often cavities develop on the permanent teeth of patients with braces (orthodontic treatment). The hypothesis is that there is no difference in the number of cavities on the permanent teeth of patients with braces compared to similar patients without braces.

DETAILED DESCRIPTION:
The purpose of this cross-sectional study is to determine the prevalence of early carious lesions (white spot lesions, or WSLs) for patients who are receiving orthodontic treatment compared to patients who are not receiving orthodontic treatment.

Subjects will be recruited from the University of Kentucky Orthodontic Clinic patient pool. Orthodontic care at the University of Kentucky College of Dentistry (UKCOD) is provided by orthodontic faculty, as well as students enrolled in the graduate orthodontic program at the UKCOD. Subjects will be invited to participate in this study after receiving an initial treatment plan with fixed appliances for at least one arch.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in this study
* Patients who receive orthodontic treatment with fixed appliances at University of Kentucky College of Dentistry
* Patients who have either metal or ceramic brackets for the treatment

Exclusion Criteria:

* Patients on a daily supplemental fluoride regimen
* Patients who has difficulty in their daily toothbrushing due to their physical disability
* Patients with lingual fixed appliances
* Patients who are pregnant
* Patients with restorations placed on the facial/buccal surface of the tooth from premolar to premolar for both arches.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants have to be 10 years older who are treatment planned for orthodontic treatment with fixed appliances in the Graduate or Faculty Orthodontic Clinic at University of Kentucky.
  Based upon the racial distribution of patients currently receiving treatment in the Graduate and Faculty Orthodontic Clinics, investigators expect that study population to be predominantly Caucasian, with minority representation from the African-American and Hispanic communities. The sample composition is expected to be equally weighted with respect to gender.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
The formation of early caries lesion on teeth (white spot lesions) | One-time assessment at participant visit (approximately 30 minutes).
  Teeth of study subjects will be evaluated for the formation of white spot lesions based on their intraoral photographs taken at their participation for the study.
The dental plaque deposit on teeth. | One-time assessment at participant visit (approximately 30 minutes).
  Teeth of study subjects will be stained with the plaque disclosing agent. After rinsing off the disclosing agent, intraoral photographs are taken for later analysis of dental plaque accumulation.
Subjects' of attitude toward the oral hygiene practice. | One-time assessment at participant visit (approximately 30 minutes).
  Participants will be asked to take an electronic questionnaire (through REDCap) consisting of 13 items that assess their dental hygiene practice and attitude toward orthodontic treatment. Individual question responses range from 0-7 (cumulative range of 0-91) with higher scores indicating more positive attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroko Nagaoka, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky College of Dentistry, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No